CLINICAL TRIAL: NCT06939751
Title: OPtimal Adult Heart Transplant Immunosuppression With MicroRNA Levels
Acronym: OPTIMAL
Status: Recruiting | Type: Observational
Sponsor: Inova Health Care Services (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: INOVA-2024-372; 1R01HL173248-01A1 (NIH)
Record Dates: First submitted 2025-04-15; First posted 2025-04-23 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2025-08

CONDITIONS: Cardiac Failure; Graft Rejection
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — Plasma and RNA
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to develop and refine a microRNA (miR) biomarker panel that can be used to phenotype net immune state after heart transplantation using circulating miRs (associated with drug doses and levels). These miRs will be used to characterize the overall immune state in adult heart transplant patients and predict patients that will go on to develop infection and rejection. MicroRNAs (miRs) are small, non-coding RNA molecules that regulate gene expression and serve as molecular biomarkers found in the circulation.

DETAILED DESCRIPTION:
The study objectives will be accomplished in a prospective, multicenter observational, longitudinal cohort study that includes ~250 Heart Transplant patients from the United States. Patients will be screened for eligibility and enrolled ~1 month (± 2 weeks) after transplant. Study participation will last 36 months.

All patients will follow the center's standard of care surveillance schedule after transplant. Blood samples will be collected for miR evaluation at:

1. specified time intervals after transplant and
2. when a clinical event of interest occurs, including treated rejection, or infection.

Research samples will be collected and used to evaluate miR expression as well as other biomarkers related to heart transplantation and immunosuppression medications. Additional data collection will include demographics, medical history, medications, human leukocyte (HLA)/donor specific antibody (DSA) evaluations, endomyocardial biopsy (EMB) echocardiography, donor-derived cell-free DNA (dd-cfDNA), and other post-transplant events and testing.

This work will form the basis for a non-invasive, genomic blood test that can be used to monitor patients after heart transplant to mitigate complications of over-immunosuppression, such as infection, without increasing the risks of under-immunosuppression, such as rejection.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years at enrollment
* Receipt of orthotopic heart transplant (OHT) within the prior 1 month ± 2 weeks
* Planned follow-up at the transplant center for a minimum of one-year.
* Patient able and willing to comply with the study visit schedule, study procedures, and study requirements.

Exclusion Criteria:

* Recipient of a multi-organ transplant
* History of prior solid organ transplant before the index heart transplant
* Ongoing mechanical circulatory support or hemodynamic instability (e.g., inotrope or vasopressor therapy)
* Ongoing need for renal replacement therapy and/or dialysis
* Active infection requiring either a) hospitalization b) treatment with antimicrobial therapy or c) reduction in immunosuppression
* Active rejection being treated with intravenous medications or plasmapheresis

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients ≥ 18 years of age from geographically and socioeconomically diverse regions of the U.S who have undergone orthotopic heart transplant (OHT)
  Patients will be screened for eligibility and enrolled within ~ 1 month after heart transplant
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2025-10-28 (Actual); Primary Completion 2031-01-01 (Estimated); Study Completion 2032-01-01 (Estimated)

PRIMARY OUTCOMES:
Time-to-Event Analysis of Circulating microRNAs (miRs) Predicting Infection in Pediatric Heart Transplant Recipients | up to 3 years post - transplant
  A time-to-event analysis will be performed to identify specific circulating microRNAs (miRs) that predict the risk of infection in heart transplant recipients. Infections are defined as any bacterial, viral, fungal, or opportunistic infection leading to: 1) hospitalization, 2) prescription of antimicrobial therapy, or 3) reduction in immunosuppression
Time-to-Event Analysis of Circulating microRNAs (miRs) Predicting Rejection in Pediatric Heart Transplant Recipients | up to 3 years post - transplant
  A time-to-event analysis will be performed to identify specific circulating microRNAs (miRs) that predict the risk of rejection in heart transplant recipients. Rejection is defined as treated rejection based on 1) endomyocardial biopsy (EMB) pathology, 2) unexplained graft dysfunction, or 3) molecular testing; leading to treatment with pulse dose steroids, monoclonal antibodies, plasmapheresis, and/or intravenous immunoglobulin (IVIg).
  EMB Pathology: Acute Cellular Rejection (ACR) Grade ≥ 2R and/or Antibody-mediated Rejection (AMR) Grade ≥ pAMR1, per International Society for Heart and Lung Transplantation (ISHLT) grading systems.
  Graft Dysfunction: Left Ventricular Ejection Fraction (LVEF) decline ≥ 10% from baseline and < 50% absolute LVEF by echocardiography.
  Molecular Testing: Presence of 2 of the following 3 criteria-presence of HLA-DSA, elevated donor-derived cell-free DNA (dd-cfDNA), or gene expression results from blood or EMB testing.

CONTACTS AND LOCATIONS:
Overall Officials: Palak Shah, MD, Principal Investigator — Inova Schar Heart and Vascular
Locations (5):
- United States (5):
  - Stanford University, Palo Alto, California
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt University, Nashville, Tennessee
  - Baylor University Medical Center, Dallas, Texas
  - Inova Health System, Falls Church, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shah P, Bristow MR, Port JD. MicroRNAs in Heart Failure, Cardiac Transplantation, and Myocardial Recovery: Biomarkers with Therapeutic Potential. Curr Heart Fail Rep. 2017 Dec;14(6):454-464. doi: 10.1007/s11897-017-0362-8. PMID 28940102
- [Background] Shah P, Agbor-Enoh S, Bagchi P, deFilippi CR, Mercado A, Diao G, Morales DJ, Shah KB, Najjar SS, Feller E, Hsu S, Rodrigo ME, Lewsey SC, Jang MK, Marboe C, Berry GJ, Khush KK, Valantine HA; GRAfT Investigators. Circulating microRNAs in cellular and antibody-mediated heart transplant rejection. J Heart Lung Transplant. 2022 Oct;41(10):1401-1413. doi: 10.1016/j.healun.2022.06.019. Epub 2022 Jun 28. PMID 35872109